CLINICAL TRIAL: NCT04517344
Title: High Flow Nasal Cannula (HFNC) Initiation Flow Rate Study - A Single Center, Randomized Controlled, Feasibility Study
Brief Title: High Flow Nasal Cannula (HFNC) Initiation Flow Rate Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol changes in the hospital
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Amy Cheng, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0816
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; HFNC; High Flow Nasal Cannula; Infants
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1, HFNC 1 L/kg/min (Experimental): The infant that is randomized to the HFNC therapy arm 1 will be placed on high flow at 1 L/kg/min (up to a maximum of 20 L/min) on fraction of inspired oxygen (FiO2) of 21 %. They will remain on FiO2 of 21% for a minimum of 10 minutes while monitoring SpO2. If oxygen saturation (SpO2) is <90%, FiO2 will be slowly increased to maintain SpO2 ≥ 90 %.
  Interventions: Other: Initial Flow Rate
- Arm 2, HFNC 1.5 L/kg/min (Experimental): The infant that is randomized to the HFNC therapy arm 2 will be placed on high flow at 1.5 L/kg/min (up to a maximum of 20 L/min) on fraction of inspired oxygen (FiO2) of 21 %. They will remain on FiO2 of 21% for a minimum of 10 minutes while monitoring SpO2. If SpO2 is <90%, FiO2 will be slowly increased to maintain SpO2 ≥ 90 %.
  Interventions: Other: Initial Flow Rate
- Arm 3, HFNC 2 L/kg/min (Experimental): The infant that is randomized to the HFNC therapy arm 3 will be placed on high flow at 2 L/kg/min (up to a maximum of 20 L/min) on fraction of inspired oxygen (FiO2) of 21 %. They will remain on FiO2 of 21% for a minimum of 10 minutes while monitoring SpO2. If SpO2 is <90%, FiO2 will be slowly increased to maintain SpO2 ≥ 90 %.
  Interventions: Other: Initial Flow Rate

INTERVENTIONS:
Other: Initial Flow Rate — Patients placed on High Flow Nasal Cannula by treating physician will be randomized to initial flow rates of 1 L/kg/min, 1.5 L/kg/min, or 2 L/kg/min

SUMMARY:
The investigators propose an open label, non-blinded, single center randomized controlled feasibility study to find the optimal initial HFNC flow rate in children less than 12 months old with clinically diagnosed moderate to severe bronchiolitis. This feasibility study is projected over December 2020 to April 2023. The study is consisted of 3 arms, comparing HFNC therapy at 1 L/kg/min, 1.5 L/kg/min, and 2 L/kg/min (20 L/min max). Moderate to severe bronchiolitis is defined clinician's assessment for the need for ICU level of care.

The primary outcome is treatment response to HFNC therapy defined by RDAI/Respiratory Assessment Change Score (RACS) ≥ 4 at 4 hours of therapy. Secondary outcome measures comprise of treatment failure requiring an escalation of care during the first 24 hours of HFNC therapy, duration of HFNC and simple nasal cannula therapy, duration of simple nasal cannula therapy, hospital and PICU length of stay (LOS), time to treatment failure, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 12 months of age
* Clinical signs of moderate to severe bronchiolitis defined by American Academy of Pediatrics
* Requires ICU level of care by clinicians' discretion
* Requiring HFNC support

Exclusion Criteria:

* Infants who required immediate need for respiratory support such as non-invasive positive pressure ventilation (NIPPV) or invasive ventilation
* Congenital heart disease,
* Immunocompromised state
* Upper airway obstruction
* Chronic lung disease
* Bronchopulmonary dysplasia,
* Home oxygen therapy requirement
* Acute trauma patients
* Baseline craniofacial malformations
* Admitted to the neonatal or cardiac ICUs
* Patients who are admitted to the floor

Ages: 7 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment response to HFNC Therapy | 4 hours of therapy
  Determined by Respiratory Distress Assessment Instrument (RDAI) score and Respiratory Assessment Change Score (RACS) and heart rate improvement by 10%.
  The RDAI score assigns a score base on respiratory rate (RR), extent of wheezing, and retractions. It ranges from 0-17, higher score indicates severe bronchiolitis.
  To determine RACS:
  * A decrease in RR by 10% is +1 change unit. Increase of 10% was defined as -1 change unit.
  * Subsequent RDAI score is subtracted from the previous RDAI score to obtain the change. (ie. if initial score is 7 and the reassessment score is 3, the patient has a score of +4) Positive score is indicative of improvement, and negative score demonstrates deterioration.
  The overall RACS is calculated as the sum of change scores. Improvement is defined as RACS ≥ 4 positive units. No improvement was defined as RACS < 4 positive units.

SECONDARY OUTCOMES:
Treatment failure to HFNC Therapy | 24 hours from time of study
  * Need for an increase in initial flow setting as determined by treating physician during the first 24 hours of hospitalization
  * Escalation to other forms of non-invasive ventilatory support (i.e. NCPAP or BIPAP)
  * Need for invasive ventilation
Length of oxygen support | 24 hours from time of study
  * Number of hours on HFNC
  * Number of hours on simple nasal cannula
Length of stay | 24 hours from time of study
  * Length of stay in the pediatric ICU
  * Length of stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cheng, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Health - Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No